CLINICAL TRIAL: NCT04474327
Title: Role of Montelukast in Modulation of Response to Sepsis in Preterm Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Hanan El-Halaby, Principal investigator, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Montelukast in neonatal sepsis
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Neonatal Sepsis
Keywords: Sepsis; Montelukast; TNF alpha; premature infant
MeSH Terms: conditions — Neonatal Sepsis; Sepsis; Premature Birth | interventions — montelukast

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Experimental): The intervention group will receive Montelukast Sodium for 10 days in addition to the conventional antibiotic therapy regimen and other supportive measures according to the policy of neonatal units and patients' needs. Montelukast sodium will be given at a dose according to body weight (1.5 kg to 2 kg, will be given 1.5 mg; greater than 2 kg, 2 mg will be given) this dose was calculated according to ( Kim et al. (2015). Four mg of the drug will be dissolved in four ml milk and 1.5 - 2 ml milk only will be given once daily at 9 pm via an orogastric tube or by oral administration for 10 days and patients of this group will be closely observed for development of Montelukast side effects as "diarrhea, colic, vomiting, fever and cough" (Adelsberg et al. 2005).
  Interventions: Drug: Montelukast Sodium
- Control group (No Intervention): The control group will receive antibiotics and other supportive measures according to the policy of neonatal units and patients' needs.

INTERVENTIONS:
Drug: Montelukast Sodium — Montelukast sodium (Singulair) will be given at a dose according to body weight. Four mg of the drug will be dissolved in four ml milk and the dose will be given once daily at 9 pm for 10 days.
  Other Names: Singulair
  Arms: Intervention group

SUMMARY:
The investigators will conduct this study to explore the role of Montelukast in treatment of neonatal sepsis and whether it has an effect on inflammatory markers, the duration of antibiotic use, or on the patients´ outcome.

DETAILED DESCRIPTION:
Since inflammatory mediators play a crucial role in the pathophysiology of sepsis so anti-inflammatory treatment, Montelukast, could be a beneficial therapy. The investigators will conduct this pilot, open-labeled, randomized controlled intervention trial on 40 newborns admitted to NICU. The study will include late preterm infants with gestational age (34 weeks to less than 37 weeks) with clinical evidence of sepsis. The study included an intervention group (n=20) that will receive oral Montelukast for 10 days with antibiotics in addition to the conventional antibiotic therapy regimen according to NICU policy while the control group (n=20) will receive antibiotics in addition to the conventional antibiotic therapy regimen according to NICU policy. After obtaining a fully informed written consent from the neonate's parents or guardians, patients will be recruited and group allocated in the study by random pick up of closed opaque sealed envelopes. Patients will be observed clinically and by laboratory investigations along the duration of hospital admission through a structured collection sheet. Demographic data, cause of admission, clinical data (vital signs, activity, feeding intolerance, respiratory symptoms, duration of oxygen support, use of inotropes) will be recorded. Blood sampling will be performed twice in both groups, on admission, and 10 days after treatment. The following investigations will be carried out: complete blood picture, C-reactive protein (CRP), tumor necrosis factor-alpha (TNF alpha), blood culture, Serum creatinine, Liver enzymes, and INR. A lumbar puncture will be performed when the treating physicians suspect meningitis. Patients in both groups will be observed along the duration of hospital admission to detect the outcome.

Patients in the intervention group, receiving Montelukast sodium (Singulair), will be given at a dose according to body weight (1.5 kg to 2 kg, will be given 1.5 mg; greater than 2 kg, will be given 2 mg). This dose was previously prescribed and given to preterm neonates suffered from bronchopulmonary dysplasia by Kim et al. (2015). Four mg of the drug will be dissolved in four ml milk and 1.5 - 2 ml milk only will be given once daily at 9 pm via an orogastric tube or by oral administration for 10 days. Along the period of NICU admission, patients receiving Montelukast will be closely observed for the development of any of its side effects that including "diarrhea, colic, vomiting, fever or cough" (Adelsberg et al., 2005).

ELIGIBILITY:
Inclusion Criteria:

* 1. Infants with gestational age from 34 weeks to less than 37 weeks (late preterm) and weighted more than 1.5 Kg with clinical evidence of neonatal sepsis (Wynn 2016).

Exclusion Criteria:

- 1. Infants presented initially with septic shock, multi-organ dysfunction syndrome (MODS), disseminated intravascular coagulopathy.

2. Infants with major congenital malformations 3. Infants with chromosomal aberrations 4. Postoperative patients.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Change in serum tumor necrosis factor (TNF) Alpha level | Measured twice: on admission and 10 days after receiving therapy
  Change in serum level of TNF alpha is assessed by the difference between the admission level and its level at 10 days after receiving the therapy.

SECONDARY OUTCOMES:
The duration of NICU admission | Counting the total duration of NICU admission
  the total duration of NICU admission
Change in serum C-reactive protein (CRP) level | Measured twice: on admission and 10 days after receiving therapy
  Serum C-reactive protein (CRP) level will be measured on admission and compare its level with the level at 10 days after receiving therapy. It will be measured in both groups
Patients improvement, deterioration (Clinically and laboratory) or death | determined at 10 days after receiving therapy
  Patients are considered 1.improved when manifested clinically by no respiratory distress, normal temperature, no oxygen support, no inotropes, alert, not lethargic, tolerate feeding, increasing in body weight and laboratory by normal CBC , normal CRP, Culture negative. 2. Partially improved if patient still on intravenous fluid therapy, still on oxygen support, still on inotropes, CRP decreasing but still positive, and CBC still abnormal. 3. Deteriorated if developed complication as coagulopathy, septic shock or MODS.
use of positive pressure ventilation and its duration | determined at 10 days after receiving therapy
  use of positive pressure ventilation (receiving mechanical ventilation or CPAP) and the duration
Duration of use of inotropes | determined at 10 days after receiving therapy
  duration of inotropes (dopamine, epinephrine, norepinephrine)

CONTACTS AND LOCATIONS:
Overall Officials: Hanan A El-Halaby, Principal Investigator — Mansoura University Children Hospital, Gomhuria street, 35116 Mansoura, Egypt
Locations (1):
- Mansoura University Childran Hospital, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] van Adelsberg J, Moy J, Wei LX, Tozzi CA, Knorr B, Reiss TF. Safety, tolerability, and exploratory efficacy of montelukast in 6- to 24-month-old patients with asthma. Curr Med Res Opin. 2005 Jun;21(6):971-9. doi: 10.1185/030079905X48456. PMID 15969897
- [Result] Kim SB, Lee JH, Lee J, Shin SH, Eun HS, Lee SM, Sohn JA, Kim HS, Choi BM, Park MS, Park KI, Namgung R, Park MS. The efficacy and safety of Montelukast sodium in the prevention of bronchopulmonary dysplasia. Korean J Pediatr. 2015 Sep;58(9):347-53. doi: 10.3345/kjp.2015.58.9.347. Epub 2015 Sep 21. PMID 26512261